CLINICAL TRIAL: NCT05245916
Title: A Phase Ia/Ib Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of IBI397 or Combination Therapies in Patients With Advanced Malignancies
Brief Title: IBI397 or Combination Therapies in Patients With Advanced Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the company's development strategy adjustment
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIBI397A101
Record Dates: First submitted 2022-01-26; First posted 2022-02-18 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IBI397 single-agent dose escalation (Experimental)
  Interventions: Drug: IBI397
- IBI397+ Rituximab (Experimental)
  Interventions: Drug: IBI397; Drug: IBI397+Rituximab
- IBI397 + Sintilimab (Experimental)
  Interventions: Drug: IBI397; Drug: IBI397+Sintilimab

INTERVENTIONS:
Drug: IBI397 — IBI397 single-agent dose escalation： Subjects will receive IBI397 until disease progression, unacceptable toxicity, withdrawal of consent, occurrence of other conditions that require discontinuation of study treatment, or the treatment duration has reached 24 months, whichever occurs first
Drug: IBI397+Sintilimab — IBI397 in combination with sintilimab： Subjects will receive IBI397 combination therapy with sintilimab until disease progression, unacceptable toxicity, withdrawal of consent, occurrence of other conditions that require discontinuation of study treatment, or the treatment duration has reached 24 months, whichever occurs first
  Arms: IBI397 + Sintilimab
Drug: IBI397+Rituximab — IBI397 in combination with rituximab： Subjects will receive IBI397 combination therapy with rituximab until disease progression, unacceptable toxicity, withdrawal of consent, occurrence of other conditions that require discontinuation of study treatment, or the treatment duration has reached 24 months, whichever occurs first
  Arms: IBI397+ Rituximab

SUMMARY:
The primary objective of this phase Ia/Ib Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of IBI397 or its Combination Therapies in Patients with Advanced Malignancies

ELIGIBILITY:
Inclusion criteria:

* Have failed the standard treatment for locally advanced, recurrent or metastatic solid tumor or have failed at least the second line standard treatment (including autologous stem cell transplantation) or have failed the first line standard treatment and are not eligible for autologous stem cell transplantation
* Willing to and able to provide written informed consent for the trial and able to comply with protocol-specified visits and related procedures
* ≥ 18 and ≤ 75 years of age on the day of signing the informed consent
* Have a performance scale of 0 or 1 on the Eastern Cooperative Oncology Group Performance Status (ECOG PS)
* Subjects with solid tumor: Have at least one measurable or assessable lesion as defined by RECIST v1.1; Subjects with lymphoma: Have at least one measurable or assessable lesion as defined by Lugano2014 criteria

Exclusion Criteria:

* Has been previously exposed to any CD47 antibody, SIRPα antibody, or CD47/SIRPα recombinant protein or other inhibitors that target the same pathway
* Is currently participating in another interventional study, except for observational (non-interventional) study or in the survival follow-up phase of an interventional study
* Requires long-term systemic hormone or any other immunosuppressive drug therapy, excluding inhaled hormone therapy
* Has acute or chronic active hepatitis B (defined as hepatitis B surface antigen [HBsAg] and/or hepatitis B core antibody positive [HBcAb] and hepatitis B virus [HBV] DNA copy number ≥ 1 × 104 copies/ml or ≥ 2000 IU/ml or higher than the lower limit of detection) or acute or chronic active hepatitis C virus (HCV) antibody positive; HCV antibody positive but RNA negative subjects are allowed
* Has a known history of severe allergic reaction to other monoclonal antibodies, or is allergic to any component of the IBI397 formulation.
* Is pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment related AEs | Up to 90 days post last dose
  Number of patients who experienced a treatment related AEs from the frist dose until 90 days after the last dose
Percentage of Subjects with Dose-Limiting Toxicities (DLTs) | Up to 28 Days following first dose
  To evaluate the safety and tolerability of IBI397 alone or in combination with Sintilimab

SECONDARY OUTCOMES:
area under the plasma concentration-time curve (AUC) | Up to 90 days post last dose
maximum concentration (Cmax) | Up to 90 days post last dose
clearance (CL) | Up to 90 days post last dose
volume of distribution (V) | Up to 90 days post last dose
half-life (t1/2) | Up to 90 days post last dose
anti-drug antibody (ADA) | Up to 90 days post last dose
  Number of Anti-Drug Antibodies (ADA) positive subjects will be counted and percentage of ADA positive subjects will be calculated to evaluate immunogenicity of IBI397
Objective response rate (ORR) | Up to 2 years after enrollment
  Objective Response Rate (ORR) is the percentage of Complete Response (CR) plus partial response (PR) assessed per RECIST v1.1 criteria for solid tumors or per Lugano2014 criteria for lymphomas

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China